CLINICAL TRIAL: NCT06706726
Title: A Prospective, Single-center, Double-arm Clinical Study to Evaluate the Effectiveness and Safety of Single-port Robotic-assisted Subcutaneous Gland Resection Combined With Immediate Breast Reconstruction in Breast Cancer
Brief Title: To Evaluate the Effectiveness and Safety of Single-port Robotic-assisted Subcutaneous Gland Resection Combined With Immediate Breast Reconstruction in Breast Cancer
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: BC-Robot-20241101
Record Dates: First submitted 2024-11-25; First posted 2024-11-27 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-11

CONDITIONS: Breast Cancer
Keywords: Single-port Robotic-assisted subcutaneous gland resection combined with immediate breast reconstruction
MeSH Terms: conditions — Breast Neoplasms | interventions — Sentinel Lymph Node Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Single-port robotic-assisted breast surgery including sentinel lymph node biopsy (Experimental): Single-port robotic-assisted（Endoscopic Instrument Control System SP1000）subcutaneous gland resection and sentinel lymph node biopsy combined with immediate breast reconstruction in the management of breast cancer
  Interventions: Procedure: sentinel lymph node biopsy
- Group B: Single-port robotic-assisted breast surgery including axillary lymph node dissection (Experimental): Single-port robotic-assisted（Endoscopic Instrument Control System SP1000）subcutaneous gland resection and axillary lymph node dissection combined with immediate breast reconstruction in the management of breast cancer
  Interventions: Procedure: Single-port robotic-assisted axillary lymph node dissection

INTERVENTIONS:
Procedure: sentinel lymph node biopsy — sentinel lymph node biopsy during the management of breast cancer
  Arms: Group A: Single-port robotic-assisted breast surgery including sentinel lymph node biopsy
Procedure: Single-port robotic-assisted axillary lymph node dissection — Single-port robotic-assisted（Endoscopic Instrument Control System SP1000) axillary lymph node dissection during the management of breast cancer
  Arms: Group B: Single-port robotic-assisted breast surgery including axillary lymph node dissection

SUMMARY:
The new technology of robotic surgery system, as an emerging technology, has shown certain application prospects in breast surgery. However, the new technology of robotic surgery system in China in the treatment of breast cancer is still in the exploratory stage and needs to be further improved. This prospective, single-center, double-arm clinical study was conducted to use the single-port robot and evaluate the effectiveness and safety of the subcutaneous gland resection combined with immediate breast reconstruction in breast cancer.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients, aged 18-75 years old; The pregnancy test (-) and reliable contraceptive methods are required for premenopausal and perimenopausal patients;
2. Patients with the diagnosed breast cancer confirmed by core needle biopsy and unilateral operation was performed; Breast cancer patients with tumor node metastasis stage 0-III according to the 8th edition of the American Joint Commission on Cancer; Preoperative clinical examination or imaging evaluation shows that the distance between the tumor and the Nipple Areolar Complex (NAC) is more than 1cm. The tumor has a diameter of 2-3 cm and can be located in any quadrant or reduced to 3 cm through preoperative neoadjuvant chemotherapy. The distance between the lesion and the skin should be at least 8-10 mm;
3. There is no clinical or imaging evidence to prove that the tumor has invaded the skin, chest wall, or nipple areola complex;
4. There are indications for breast preservation, but the patient has a strong desire for reconstruction and is unwilling to undergo breast preservation surgery;
5. Preventive mastectomy (BRCA1/2 malignant mutation with obvious family history of breast cancer and other high-risk groups);
6. Preoperative clinical manifestations and imaging data showed no distant metastasis;
7. No history of breast cancer or other serious underlying diseases in the past;
8. Karnofsky performance status score ≥ 70;
9. Eastern Cooperative Oncology Group score ≤ 2 ;
10. The surgical procedure includes a single-port robot (Endoscopic Instrument Control System SP1000) for subcutaneous gland resection, sentinel lymph node biopsy, axillary lymph node dissection and immediate breast reconstruction;
11. Participants are able to understand the research process, voluntarily join the study, sign informed consent forms, have good compliance, and cooperate with follow-up;
12. No swallowing difficulties; No shoulder joint movement disorders;
13. Complete clinical data.

Exclusion Criteria:

1. Male breast cancer or inflammatory breast cancer;
2. Metastatic breast cancer (stage IV); Tumor invasion of the skin, pectoralis major muscle, or NAC;
3. The clinical data is basically incomplete;
4. Previously received chemotherapy in an external hospital or has undergone tumor resection in an external hospital;
5. Bilateral breast cancer surgery;
6. Other surgical methods;
7. Preoperative distant metastasis or supraclavicular lymph node dissection;
8. Complicated with other malignant tumors or had malignant tumors other than breast cancer in recent 5 years;
9. The serious disease of non malignant tumors combined will affect the patient's compliance or put the patient in a dangerous state;
10. Dementia, intellectual disability, or any mental illness that hinders understanding of informed consent forms.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-12-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Local recurrence free survival rate | Ten years
  Local recurrence refers to the recurrence of the chest wall or breast on the same side as the surgical site.

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol